CLINICAL TRIAL: NCT04317274
Title: Online Trial Examining Validity of the Shared Decision Making Process Survey With Video Vignettes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: University of Massachusetts, Boston (Other)
Responsible Party: Principal Investigator, Karen Sepucha, Director of the Health Decision Sciences Center, Massachusetts General Hospital
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Other
Other Study IDs: 2019P001434
Record Dates: First submitted 2020-03-17; First posted 2020-03-23 (Actual); Results first posted 2024-01-05 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2023-03

CONDITIONS: Colorectal Cancer; High Cholesterol
MeSH Terms: conditions — Colorectal Neoplasms; Hypercholesterolemia

STUDY DESIGN:
Intervention Model Description: Subjects were randomly assigned to one of the two clinical conditions (colorectal cancer screening or high cholesterol) then randomly assigned to view the two videos in one of two orders. Participants either viewed the good shared decision making video first (and the poor shared decision making video second) or the poor shared decision making video first (and the good shared decision making video second). Thus we used a 2 (clinical condition; colorectal cancer screening v. high cholesterol) x 2 (video; good v. poor) x 2 (order; good first v. poor first) factorial design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- High Cholesterol Good Video First (Experimental): Participants see videos of a conversation around taking medications (statins) for high cholesterol. Patients see good video first and poor video second.
  Interventions: Behavioral: Good high cholesterol video; Behavioral: Poor high cholesterol video
- Colorectal Cancer Good Video First (Experimental): Participants see videos of a conversation around screening for colorectal cancer. Patients see good video first and poor video second.
  Interventions: Behavioral: Good colon cancer screening video; Behavioral: Poor colon cancer screening video
- High Cholesterol Poor Video First (Experimental): Participants see videos of a conversation around taking medications (statins) for high cholesterol. Patients see poor video first and good video second.
  Interventions: Behavioral: Good high cholesterol video; Behavioral: Poor high cholesterol video
- Colorectal Cancer Poor Video First (Experimental): Participants see videos of a conversation around screening for colorectal cancer. Patients see poor video first and good video second.
  Interventions: Behavioral: Good colon cancer screening video; Behavioral: Poor colon cancer screening video

INTERVENTIONS:
Behavioral: Good high cholesterol video — The short video illustrated key components of a high quality shared decision making conversation between a doctor and patient actor around treatment of high cholesterol.
  Arms: High Cholesterol Good Video First; High Cholesterol Poor Video First
Behavioral: Poor high cholesterol video — The short video illustrated a typical conversation between a doctor and patient actor that did not cover key aspects of share decision making around treatment of high cholesterol.
  Arms: High Cholesterol Good Video First; High Cholesterol Poor Video First
Behavioral: Good colon cancer screening video — The short video illustrated key components of a high quality shared decision making conversation between a doctor and patient actor around screening for colorectal cancer.
  Arms: Colorectal Cancer Good Video First; Colorectal Cancer Poor Video First
Behavioral: Poor colon cancer screening video — The short video illustrated a typical conversation between a doctor and patient actor that did not cover key aspects of share decision making around screening for colorectal cancer.
  Arms: Colorectal Cancer Good Video First; Colorectal Cancer Poor Video First

SUMMARY:
This study will recruit subjects online and randomly assigned them to one of four arms. The arms vary by clinical decision (colorectal cancer screening or treatment of high cholesterol) by video order (poor shared decision making followed by good or good shared decision making followed by poor). Participants will view two videos and complete the Shared Decision Making process survey along with a few other measures after each video. Our main hypothesis is that respondents watching the good shared decision making videos will score higher on the Shared Decision Making Process survey compared to those watching the poor videos.

DETAILED DESCRIPTION:
Study staff are working with a national sampling firm to recruit subjects and obtain 400 responses. Subjects were randomly assigned to one of four arms. (1) Colorectal cancer screening good shared decision making video then poor video second (2) Colorectal cancer screening poor shared decision making video then good video (3) Treatment of high cholesterol good video then poor video and (4) Treatment of high cholesterol poor shared decision making video first then good video. Participants completed measures of Shared Decision Making after each video.

The sample size was determined to ensure sufficient power to detect differences between the good and the poor shared decision making videos in this repeated measure design and analyses were planned to be separate for each arm (i.e. one analysis for the colorectal cancer screening videos and a separate parallel analysis of the statins for high cholesterol video). To detect an eta2 effect size of .04 with an alpha of 0.05 with 80% power would require 190 observations per clinical condition. Study staff rounded this to 200 observations per clinical condition, for a total required sample size of 400 patients.

The interventions were short Shared Decision Making Videos that were developed as part of two training courses on shared decision making by investigators at Massachusetts General Hospital.

For the analyses, study staff will examine the descriptives of the Shared Decision Making Process items for the two clinical conditions and orders. Study staff will examine rates of missing data to determine acceptability, and will examine descriptive results to see whether the scores span the range of total possible scores, are normally distributed, and whether there is evidence of floor or ceiling effects. Then, study staff examine discriminant validity of the measure by examining whether scores for the good videos are higher then for the poor videos. Further, study staff will examine concurrent validity with the alternative shared decision making measure.

ELIGIBILITY:
Inclusion Criteria:

* Speak English
* No prior diagnosis of colorectal cancer
* No history of heart attack
* No history of stroke

Exclusion Criteria:

* None

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 401 (Actual)
Dates: Start 2020-03-13 (Actual); Primary Completion 2020-04-08 (Actual); Study Completion 2020-04-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen Sepucha, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The study team will create a complete, cleaned, de-identified copy of the final data set for each online field test. After the main analyses have been published, information for accessing the data will be made available on the Health Decision Sciences Center website and in publications of the data. Dr. Sepucha will share a de-identified data set with outside investigators at no cost, according to approved Massachusetts General Hospital/Partners policies for data sharing. Investigators from other sites will be able to request the data and will be required to complete a data use agreement that ensures that all local Institutional Review Board requirements are met before using the data, that they will not attempt to identify any data in the dataset, and that they will not share the data set with anyone outside their project team.
Supporting Information: Study Protocol, SAP, Analytic Code

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | High Cholesterol Good Video First | Colorectal Cancer Good Video First | High Cholesterol Poor Video First | Colorectal Cancer Poor Video First
Started | 97 | 94 | 103 | 107
Completed | 95 | 91 | 99 | 103
Not Completed | 2 | 3 | 4 | 4
Not completed — participant did not provide enough information to calculate a shared decision making process score | 2 | 3 | 4 | 4

BASELINE CHARACTERISTICS:
Population: Participants who provided sufficient information to calculate the shared decision making process score (primary outcome of interest)
Groups:
- Total: Total of all reporting groups
Arm/Group | High Cholesterol Good Video First | Colorectal Cancer Good Video First | High Cholesterol Poor Video First | Colorectal Cancer Poor Video First | Total
Number analyzed (Participants) | 95 | 91 | 99 | 103 | 388
Age, Continuous [Mean (Standard Deviation); unit: years] | 45 (16) | 45 (16) | 45 (16) | 44 (16) | 45 (16)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 66 | 64 | 72 | 67 | 269
  Male | 28 | 27 | 26 | 36 | 117
  Genderfluid | 1 | 0 | 0 | 0 | 1
  Nonbinary | 0 | 0 | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 4 | 10 | 11 | 35
  Not Hispanic or Latino | 85 | 87 | 89 | 92 | 353
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 1 | 1 | 5
  Asian | 5 | 6 | 6 | 9 | 26
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 0 | 0 | 2
  Black or African American | 15 | 12 | 11 | 12 | 50
  White | 65 | 65 | 70 | 75 | 275
  More than one race | 1 | 2 | 3 | 1 | 7
  Unknown or Not Reported | 6 | 4 | 8 | 5 | 23
Region of Enrollment [Number; unit: participants]
  United States | 95 | 91 | 99 | 103 | 388

OUTCOME MEASURES:

1. Primary Outcome: Shared Decision Making Process Score
Description: The Shared Decision Making Process is a short, 4-item patient-reported survey that measures the amount of shared decision making that occurs in an interaction. Scores range from 0-4 where higher values indicate a better shared decision making process occurred.
Time Frame: Immediately after viewing each video (typically within 15 minutes of watching the video)
Population: participants who answered the shared decision making process items and provided sufficient information to calculate a SDM Process score.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | High Cholesterol Good Video First | Colorectal Cancer Good Video First | High Cholesterol Poor Video First | Colorectal Cancer Poor Video First
Number analyzed (Participants) | 95 | 91 | 99 | 103
score on a scale
  Poor video score | 2.62 (1.02) | 1.82 (1.30) | 2.55 (1.01) | 2.06 (1.1)
  Good video score | 3.36 (0.61) | 3.08 (0.75) | 3.10 (0.79) | 3.29 (0.66)
Statistical Analysis 1: Comparison: High Cholesterol Good Video First vs High Cholesterol Poor Video First; We tested for interaction effect of order and video version within the high cholesterol group; Test type: Other; p = 0.21, Mixed Models Analysis; Note: original plan was to conduct ANOVAs, but failed tests of assumptions; Slope = -0.19
Statistical Analysis 2: Comparison: Colorectal Cancer Good Video First vs Colorectal Cancer Poor Video First; We tested for interaction effect of order and video version within the colorectal cancer group; Test type: Other; p < 0.001, Mixed Models Analysis; Original plan was to conduct ANOVAs, but failed tests of assumptions; Slope = -1.23

2. Secondary Outcome: Shared Decision Making Questionnaire (SDM-Q-9)
Description: The SDM-Q9 is a 9-item patient reported measure of the amount of shared decision making that occurs in an interaction. Items are scored on a six-point Likert scale from 0 (completely disagree) to 5 (completely agree); items are summed up to a total raw score between 0-45. The score is then transformed to range from 0-100 where higher values indicate a better shared decision making process occurred.
Time Frame: Immediately after viewing each video (typically within 15 minutes of watching the video)
Population: Participants who completed the 9-item SDM-Q9 measure. 388/388 participants provided sufficient information to calculate an SDMQ9 score.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | High Cholesterol Good Video First | Colorectal Cancer Good Video First | High Cholesterol Poor Video First | Colorectal Cancer Poor Video First
Number analyzed (Participants) | 95 | 91 | 99 | 103
score on a scale
  Poor video score | 70.72 (19.72) | 49.69 (27.06) | 65.13 (16.48) | 55.73 (22.85)
  Good video score | 82.11 (14.42) | 80.31 (18.33) | 80.89 (16.47) | 84.96 (15.22)
Statistical Analysis 1: Comparison: High Cholesterol Good Video First vs High Cholesterol Poor Video First; We examined the correlation between SDM Process and SDM-Q9 scores in the high cholesterol group; Test type: Other; p < .001, Pearson's correlation coefficient; Slope = 0.58
Statistical Analysis 2: Comparison: Colorectal Cancer Good Video First vs Colorectal Cancer Poor Video First; We examined the correlation between SDM Process and SDM-Q9 scores in the colorectal cancer group; Test type: Other; p < .001, Pearson's correlation coefficient]; Slope = 0.71

3. Secondary Outcome: Healthcare Provider Treatment Recommendation
Description: Single item asking what the healthcare provider recommended the patient do in the video
Time Frame: Immediately after viewing each video (typically within 15 minutes of watching the video)
Population: Participants who answered the healthcare provider recommendation question. 388/388 provided sufficient information for this outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | High Cholesterol Good Video First | Colorectal Cancer Good Video First | High Cholesterol Poor Video First | Colorectal Cancer Poor Video First
Number analyzed (Participants) | 95 | 91 | 99 | 103
Participants
  Poor Video responses: Take medicine | 80 | NA — response option only administered to high cholesterol group | 74 | NA — response option only administered to high cholesterol group
  Poor Video responses: Have a colonoscopy | NA — response option only administered to colorectal cancer screening group | 60 | NA — response option only administered to colorectal cancer screening group | 77
  Poor Video responses: Do a stool-based test | NA — response option only administered to colorectal cancer screening group | 13 | NA — response option only administered to colorectal cancer screening group | 6
  Poor Video responses: Not take medicine/Not be screened | 2 | 2 | 3 | 1
  Poor Video responses: Do something else | 1 | 2 | 3 | 1
  Poor Video responses: Did not express an opinion | 12 | 14 | 19 | 18
  Good video responses: Take medicine | 61 | NA — response option only administered to high cholesterol group | 64 | NA — response option only administered to high cholesterol group
  Good video responses: Have a colonoscopy | NA — response option only administered to colorectal cancer screening group | 22 | NA — response option only administered to colorectal cancer screening group | 22
  Good video responses: Do a stool-based test | NA — response option only administered to colorectal cancer screening group | 41 | NA — response option only administered to colorectal cancer screening group | 57
  Good video responses: Not take medicine/Not be screened | 3 | 0 | 7 | 1
  Good video responses: Do something else | 7 | 0 | 7 | 1
  Good video responses: Did not express an opinion | 24 | 28 | 21 | 22

4. Secondary Outcome: Patient Treatment Preference
Description: Single item asking what the patient in the video wanted to do
Time Frame: Immediately after viewing each video (typically within 15 minutes of watching the video)
Population: Participants who answered the patient treatment preference question. Only 385/388 provided sufficient information for this outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | High Cholesterol Good Video First | Colorectal Cancer Good Video First | High Cholesterol Poor Video First | Colorectal Cancer Poor Video First
Number analyzed (Participants) | 95 | 90 | 99 | 101
Participants
  Poor video scores: Take medicine | 25 | NA — response option only administered to high cholesterol group | 25 | NA — response option only administered to high cholesterol group
  Poor video scores: Have a colonoscopy | NA — response option only administered to colorectal cancer screening group | 15 | NA — response option only administered to colorectal cancer screening group | 8
  Poor video scores: Do a stool-based test | NA — response option only administered to colorectal cancer screening group | 19 | NA — response option only administered to colorectal cancer screening group | 20
  Poor video scores: Not take medicine/Not be screened | 55 | 53 | 44 | 67
  Poor video scores: Do something else | 15 | 3 | 30 | 6
  Poor video scores: Missing | 0 | 0 | 0 | 0
  Good video scores: Take medicine | 31 | NA — response option only administered to high cholesterol group | 54 | NA — response option only administered to high cholesterol group
  Good video scores: Have a colonoscopy | NA — response option only administered to colorectal cancer screening group | 19 | NA — response option only administered to colorectal cancer screening group | 8
  Good video scores: Do a stool-based test | NA — response option only administered to colorectal cancer screening group | 60 | NA — response option only administered to colorectal cancer screening group | 87
  Good video scores: Not take medicine/Not be screened | 45 | 10 | 21 | 6
  Good video scores: Do something else | 19 | 1 | 23 | 0
  Good video scores: Missing | 0 | 0 | 1 | 0

5. Secondary Outcome: Adapted Controlled Preference Item
Description: Single item asking the participant who made the ultimate decision in the video. The categorical response options are 1) the patient made the decision, 2)the provider made the decision, or 3) both patient and provider made the decision together.
Time Frame: Immediately after viewing each video (typically within 15 minutes of watching the video)
Population: Participants who completed the adapted controlled preference question. 388/388 participants provided sufficient information for this outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | High Cholesterol Good Video First | Colorectal Cancer Good Video First | High Cholesterol Poor Video First | Colorectal Cancer Poor Video First
Number analyzed (Participants) | 95 | 91 | 99 | 103
Participants
  Poor video responses: Mainly the doctor | 50 | 49 | 51 | 59
  Poor video responses: Mainly the patient | 11 | 18 | 16 | 11
  Poor video responses: The doctor and the patient made the decision together | 34 | 24 | 31 | 33
  Poor video responses: Missing | 0 | 0 | 1 | 0
  Good video responses: Mainly the doctor | 16 | 16 | 16 | 11
  Good video responses: Mainly the patient | 24 | 35 | 28 | 37
  Good video responses: The doctor and the patient made the decision together | 54 | 40 | 55 | 55
  Good video responses: Missing | 1 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Survey responses were assessed within 2 weeks of survey completion for evidence of adverse events.
Description: Participants had the contact information for 3 members of the study team to contact with any problems or to report any adverse events. Of note, this was not a cross-over study, participants were selected for 1 of 2 topics (colorectal cancer screening or high cholesterol) and then randomized to viewing order to create 4 arms. Each participant in the listed arms saw both videos in the same order and were combined for assessment of adverse events.
Arm/Group | High Cholesterol Good Video First | Colorectal Cancer Good Video First | High Cholesterol Poor Video First | Colorectal Cancer Poor Video First
All-Cause Mortality (participants affected / at risk) | 0/97 | 0/94 | 0/103 | 0/107
Serious Adverse Events (participants affected / at risk) | 0/97 | 0/94 | 0/103 | 0/107
Other Adverse Events (participants affected / at risk) | 0/97 | 0/94 | 0/103 | 0/107

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-03-06): https://cdn.clinicaltrials.gov/large-docs/74/NCT04317274/Prot_SAP_000.pdf